CLINICAL TRIAL: NCT01003028
Title: Reduction of Remifentanil-related Complications by Limiting Maximum Plasma Concentration During Target-controlled Infusion
Brief Title: Reduction of Remifentanil-related Complications
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CW Jung_TCI_Remi_Cpmax
Record Dates: First submitted 2009-10-23; First posted 2009-10-28 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia
Keywords: Total intravenous anesthesia; Maximum plasma concentration of remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited (Experimental): Limit the maximum plasma concentration target to 9.8 ng/ml
  Interventions: Drug: Remifentanil (Limited) - Target Controlled Infusion system
- Control (Active Comparator): Use 20 ng/ml as max plasma concentration
  Interventions: Drug: Remifentanil (Control) - Target Controlled Infusion system

INTERVENTIONS:
Drug: Remifentanil (Limited) - Target Controlled Infusion system — Limit max plasma concentration to 9.8 ng/ml
  Arms: Limited
Drug: Remifentanil (Control) - Target Controlled Infusion system — Use 20 ng/ml as max plasma concentration
  Arms: Control

SUMMARY:
This study is intended to evaluate the effect of decreasing the maximum plasma concentration target of remifentanil of the Target Controlled Infusion system on the the incidence of major and minor side-effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 year old
* ASA class 1-3 scheduled for elective surgery

Exclusion Criteria:

* history of neurologic or mental disorder
* uncontrolled pulmonary or cardiovascular disease
* history of adverse reactions to opioids
* history of drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
hypotension more than 25% from baseline | during remifentanil loading

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea